CLINICAL TRIAL: NCT01293279
Title: HCV Viral Genotyping Distribution and Genetic Variation in IL28B Distributions Among the Han Ethnic Chinese in China
Brief Title: HCV (Hepatitis C Virus) Viral and Host Genotyping (IL28B, Interleukin 28B) in China
Acronym: HCV
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Lai Wei, Professor, Peking University People's Hospital
Other Study IDs: CCgenos
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-06

CONDITIONS: Hepatitis C
Keywords: HCV viral genotypes; host genotypes; IL28B; ITPA; RNA; China
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — By having the approvals from the EC and China National Human Genetic Resource Management Office (under China Ministry of Health) and having the patient informed consent, blood samples of all recruited patients will be retained under the proper conditions in Peking University People's Hospital, Beijing, China
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HCV Patients who are treatment naive: Han ethnic Chinese male or female ≥ 18 years old with recent a confirmation of anti-HCV-antibody positive and HCV RNA positive but antiviral or interferon treatment naive at the time this study starts from 28 university affiliated hospital throughout China.

SUMMARY:
The primary objective of this study is to estimate the distributions of HCV viral/human genotypes (including IL28B and inosine triphosphatase, ITPA), and HCV RNA level among ITPA gene among 1000 Han ethnic Chinese patients with HCV who are antiviral treatment naive at the time the study is conducted.

DETAILED DESCRIPTION:
A sample of 1000 Han ethnic Chinese male or female who are ≥ 18 years old with a recent confirmation of anti-HCV-antibody positive and HCV RNA positive but antiviral treatment naive from 28 university affiliated hospital in China. The primary objective of this study is to estimate the distributions of HCV Viral genotyping(ie, genotype 1 through 6 and their known subtypes), and host genotypes, both inosine triphosphatase (ITPA) gene, and IL28B. This study also collects other data including patients' demographic and clinical characteristics. There is no active antiviral treatments and no follow-up in this study.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* Han ethnic
* ≥ 18 years old
* recent confirmation of anti-HCV-antibody positive and HCV RNA positive 30 days prior to the recruitment
* antiviral or interferon treatment naive

Exclusion Criteria:

* < 18 years old
* not Han ethnic
* treated by antiviral before this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000 Han ethnic Chinese in China
Sampling Method: Probability Sample
Enrollment: 997 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Hepatitis C viral and host genotypes | Confirmation of an HCV infection 30 days prior to the recruitment
  To describe the distributions of both HCV viral and host genotypes (IL28B and ITPA) among antiviral treatment naive HCV patients

SECONDARY OUTCOMES:
Hepatitis C RNA levels | Confirmation of an HCV infection 30 days prior to the recruitment
  To describe the distribution of HCV RNA levels in antiviral treatment-naive HCV patients

CONTACTS AND LOCATIONS:
Overall Officials: Lai Wei, MD, Principal Investigator — Peking University People's Hospital, Peking University Hepatology Institute; Hong Li, Ph.D., MPH, Study Director — Bristol-Myers Squibb
Locations (1):
- Lai Wei, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wu N, Rao HY, Yang WB, Gao ZL, Yang RF, Fei R, Gao YH, Jin Q, Wei L. Impact of hepatitis C virus genotype 3 on liver disease progression in a Chinese national cohort. Chin Med J (Engl). 2020 Feb 5;133(3):253-261. doi: 10.1097/CM9.0000000000000629. PMID 31934936
- [Derived] Huang R, Rao H, Shang J, Chen H, Li J, Xie Q, Gao Z, Wang L, Wei J, Jiang J, Sun J, Jiang J, Wei L. A cross-sectional assessment of health-related quality of life in Chinese patients with chronic hepatitis c virus infection with EQ-5D. Health Qual Life Outcomes. 2018 Jun 15;16(1):124. doi: 10.1186/s12955-018-0941-8. PMID 29903024
- [Derived] Yan LB, Rao HY, Ma YJ, Bai L, Chen EQ, Du LY, Yang RF, Wei L, Tang H; CCgenos Study Group. Hepatitis B virus infection in Chinese patients with hepatitis C virus infection: prevalence, clinical characteristics, viral interactions and host genotypes: a nationwide cross-sectional study. BMJ Open. 2016 Oct 12;6(10):e012016. doi: 10.1136/bmjopen-2016-012016. PMID 27733412